CLINICAL TRIAL: NCT04252989
Title: Atropine 0.01% Eyedrops for Evolutive Myopia Treatment in Children. MYOPSTOP
Brief Title: Atropine 0.01% Eyedrops for Evolutive Myopia Treatment in Children
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN962019/CHUSTE
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Myopia; Children
Keywords: atropine
MeSH Terms: conditions — Myopia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with active myopia treated with ATROPINE eye drops
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — * Demographic data: age, sex
  * Ophthalmological history: refraction of parents, previous refractions
  * Ophthalmological data at each examination: intra-ocular pression, objective refraction after "fog", cycloplegia with SKIACOL, slit lamp, dilated eye exam, biometrics
  * Potential undesirable events (halos, photophobia...)

SUMMARY:
Prevalence of myopia and its complications has been increasing over the past decades, especially among children and adolescents. It reaches record levels in Asia: nearly 80% of the population in some regions in 2012 where the investigators speak in terms of epidemic.

ATROPINE 0.01% eyedrops one drop per day is today an evolutive myopia treatment, whose results are promising.

The investigators use this eye drops in our clinical practice at hospital of Saint-Etienne since 2017.

Few clinical data have been published so far concerning the French population.

The investigators would like to build a database so that the investigators can publish our results and share our experience.

ELIGIBILITY:
Inclusion Criteria:

* Children with active myopia treated with ATROPINE 0.01% eye drops
* patient affiliated with a social security organization
* agreement of both parents

Exclusion Criteria:

* non compliance with treatment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with active myopia treated with ATROPINE 0.01% eye drops
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
previous refractions | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice
refraction of parents | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice
intra-ocular pression | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice
objective refraction after "fog" | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice
cycloplegia with SKIACOL | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice
slit lamp | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice
dilated eye exam | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice
biometrics | every 6 months up to age 18 years
  effectiveness of ATROPINE 0.01% eyedrops in our current clinical practice

SECONDARY OUTCOMES:
undesirable events collection | every 6 months up to age 18 years
  measured the tolerance of ATROPINE 0.01% eyedrops. Number of participants with treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Caroline TRONE, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No